CLINICAL TRIAL: NCT03167580
Title: REstricted Versus Liberal Positive End-Expiratory Pressure in Patients Without Acute Respiratory Distress Syndrome
Brief Title: REstricted Versus Liberal Positive End-Expiratory Pressure in Patients Without ARDS
Acronym: RELAx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amphia Hospital (Other); Gelre Hospitals (Other); Isala (Other); Maastricht University Medical Center (Other); Medical Center Haaglanden (Other); Onze Lieve Vrouwe Gasthuis (Other); St. Antonius Hospital (Other); Amsterdam UMC, location VUmc (Other); Dijklander Ziekenhuis (Other); Spaarne Gasthuis (Other); HagaZiekenhuis (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr. Marcus J. Schultz, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELAx
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Ventilator-free Days

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilation with restricted PEEP level (Experimental): Use of the restricted PEEP level (0 - 5 cm H2O, the lowest possible PEEP level) after intubation and during all mechanical ventilation.
  Interventions: Procedure: restricted PEEP
- Ventilation with liberal PEEP Level (Active Comparator): Use of the liberal PEEP level (8 cm H2O) after intubation and during all mechanical ventilation.
  Interventions: Procedure: liberal PEEP

INTERVENTIONS:
Procedure: restricted PEEP — Patients are randomized and ventilated with restricted PEEP (the lowest possible PEEP level, 0 - 5 cm H2O)
  Arms: Ventilation with restricted PEEP level
Procedure: liberal PEEP — Patients are randomized and ventilated with liberal PEEP (the median PEEP level used in the Netherlands, 8 cm H2O)
  Arms: Ventilation with liberal PEEP Level

SUMMARY:
The 'REstricted versus Liberal positive end-expiratory pressure in patients without Acute respiratory distress syndrome' (RELAx) trial is a national multicenter, open randomized controlled trial in ICU patients without ARDS at start of ventilation. It will be the first RCT comparing ventilation with the lowest possible positive end-expiratory pressure (PEEP) level with ventilation with the median PEEP level currently practiced in the Netherlands that recruits a sufficient number of patients to test the hypothesis that ventilation with the lowest possible PEEP level is non-inferior to ventilation with a PEEP level of 8 cm H2O with regard to objective and patient-relevant clinical endpoints.

DETAILED DESCRIPTION:
Research question:

Is mechanical ventilation with the lowest possible PEEP level, as compared to mechanical ventilation with the PEEP level currently practiced, non inferior in terms of the number of ventilator-free days at days 28 in patients without ARDS?

Study design:

National multicenter, non-inferiority, open randomized controlled trial in intubated and ventilated adult ICU patients without ARDS.

Centers:

13 centers in The Netherlands will participate in this trial:

* Academic Medical Center, University of Amsterdam
* Amphia Hospital, Breda
* Gelre Hospitals, Apeldoorn
* HagaZiekenhuis, Den Haag
* Isala Clinics, Zwolle
* Maastricht University Medical Center, Maastricht
* Haaglanden Medical Center, Den Haag
* Onze Lieve Vrouwe Gasthuis, Amsterdam
* Rijnstate Hospital, Arnhem
* Spaarne Gasthuis, Hoofddorp and Hoofddorp
* Sint Antonius Hospital, Nieuwegein
* VU Medical Center, Amsterdam
* Westfriesgasthuis, Hoorn

Monitoring:

Monitoring of patients safety and reviewing of safety issues is performed by a designated independent Data Safety and Monitoring Board (DSMB).The DSMB watches over the ethics of conducting the study in accordance with the Declaration of Helsinki.

Study population:

Adult intensive care unit(ICU) patients without ARDS with an anticipated duration of ventilation of at least 24 hours, within 1 hour after initiation or admittance to the ICU if already intubated and ventilated admission.

Sample Size Calculation:

Group size calculation is focused on demonstrating non-inferiority. When the sample size in each is 445, an one-sided non-inferiority t-test (targeted at 0.05 significance level) for the difference in means of log-transformed normalized data has a 80% power to reject the null hypothesis that the number of VFD-28 in the 'restricted PEEP'-arm is inferior to the number of VFD-28 in the 'liberal PEEP'-arm by a margin of 10% anticipating on a coefficient of a variation of 0.70 (www.stichting-nice.nl), in favor or the alternative hypothesis that the number of VFD-28 in the 'restricted PEEP'-arm is non-inferior.

The choice for a margin of 10% is motivated by what is considered acceptable from a clinical point of view as the maximal acceptable reduction of the ventilator-free period for non-inferiority. Clinically this margin means that an increase of > 10% in the duration of mechanical ventilation will reduce the VFD-28 with > 12 hours (calculated over the expected mean duration of mechanical ventilation of 5 days) (www.stichting-nice.nl), which will be considered inferior. To allow for an anticipated drop out of 10% a total of 980 patients will be included.

Methods:

Patients in participating intensive care units (ICU) are screened for eligibility and randomized within one hour of initiation of invasive ventilation or, if already intubated and ventilated before admission, on ICU admission. Demographic data on screened patients regardless of meeting enrollment criteria will be recorded (registry: age, gender, type of surgery).

Randomization will be performed using a dedicated, password protected, SSL-encrypted website. Randomization sequence is generated by a dedicated computer randomization software program. Due to the nature of the intervention, blinding is not possible.

Patients are randomly assigned in a 1:1 ratio to the 'restricted PEEP'-arm (i.e. lowest possible PEEP level, 0-5 cm H2O) or to the 'liberal PEEP'-arm (i.e. a PEEP level of 8 cm H2O, the median PEEP level applied in the Netherlands)

The allowed ventilation modes are: volume-controlled or pressure-controlled ventilation, and pressure support ventilation. Automated modes, in particular those that automatically change PEEP and FiO2, are never allowed. With volume-controlled and pressure-controlled ventilation the inspiration-to-expiration ratio is set at 1:2. With volume-controlled ventilation the inspiration time and pause are set at 25% and 10%, respectively. With pressure support ventilation the highest possible pressure rise is chosen, and cycling off is set at 25%. Tidal volume size is between 6-8 ml/kg predicted body weight, which is calculated according to the following formula 50 + 0.91 x (centimeters of height - 152.4) for males and 45.5 + 0.91 x (centimeters of height - 152.4) for females. The respiratory rate is adjusted to obtain a normal arterial blood pH (7.35 to 7.45). In case of metabolic acidosis or alkalosis, a lower or higher than normal PaCO2 can be accepted, which is left to the discretion of the attending physician. Recruitment maneuvers are allowed when deemed necessary, but the decision to perform a recruitment maneuver is also left to the discretion of the attending physician.

- Patients randomized to the 'restricted PEEP'-arm start with a PEEP level of 5 cm H2O and with an inspired oxygen fraction (FiO2) between 0.21 and 0.6. The goal is to ventilate with the lowest possible PEEP level resulting in an acceptable level of oxygenation. For this, the operator, usually the attending ICU nurse, will reduce the level of PEEP in steps of 1 cm H2O to a minimum level of 0 cm H2O. Every 15 minutes the PEEP level is reduced with 1 cm H2O, as long as the pulse oximetry reading shows a SpO2 > 92% or the arterial blood gas shows a PaO2 > 8 kPa. Thereafter, ventilation continues with the lowest PEEP level at which the SpO2 > 92% or PaO2 > 8 kPa, using a FiO2 of between 0.21 and 0.6. In case the SpO2 drops below 92% or the PaO2 drops below 8 kPa, brief periods up to 5 minutes may be tolerated, first FiO2 is increased up to maximum 0.6 before PEEP is increased in steps of 1 cm H2O until 5 cm H2O.

These so-called down-titrations of the PEEP level are allowed as often as wanted, but with a minimum of three per ICU nurse shift.

Patients are weaned from the ventilator and tracheally extubated using the lowest PEEP level.

- Patients randomized to the 'liberal PEEP'-arm start with a PEEP level of 8 cm H2O and with a FiO2 between 0.21 and 0.6. The goal is to ventilate the patient mainly at this level of PEEP till tracheal extubation. For this, the operator will increase the level of PEEP, if a level of < 8 cm H2O was used, to 8 cm H2O in one single step. Thereafter, ventilation continues at 8 cm H2O using a FiO2 of between 0.21 and 0.6. In case the SpO2 drops below 92% or the PaO2 drops below 8 kPa, first FiO2 is increased to maximum 0.6 before the level of PEEP is further increased.

Patients are weaned of the ventilator and tracheally extubated using a PEEP level of 8 cm H2O. If preferred, the level of PEEP can be set at 5 cm H2O for one to two hours directly before tracheal extubation, left to the discretion of the attending physician.

- The oxygenation target ranges for SpO2 and PaO2 are 92% to 96%, and 8 kPa to 11.5 kPa, respectively. Oxygenation will be maintained in the target ranges primarily by adjusting the FiO2, which is typically set between 0.21 and 0.6 to maintain the oxygenation target ranges. The oxygenation target is primarily assessed by peripheral saturation (SpO2) as measured by pulse oximetry and only in case of unreliable reading the oxygenation will be assessed by the arterial blood oxygen pressure (PaO2).

For patients in whom the risk of severe hypoxemia could be become unacceptable during the trial (e.g., in patients who develop: ongoing cardiac ischemia due to cardiac infarction and failed revascularization, delayed cerebral ischemia after subarachnoid hemorrhage, increased and uncontrollable intracranial pressure (of ≥ 18 mmHg), necrotizing fasciitis or severe untreatable anemia such as with Jehovah's Witnesses), the target ranges for oxygenation can be increased to SpO2 and PaO2 of 94% to 96%, and 9 kPa to 11.5 kPa, respectively.

- In all patients who receive assist ventilation, three times a day it should be tested whether the patient accepts assisted ventilation; this should also be tried when a patient shows respiratory muscle activity during assist ventilation.

The attending physician decides when to tracheally extubate a patient, based on general extubation criteria (i.e. responsive and cooperative, adequate cough reflex, adequate oxygenation with FiO2 ≤ 0.4, hemodynamically stable, no uncontrolled arrhythmia and a rectal temperature > 36 Celsius and after successfully passing a spontaneous breathing trial (SBT) with a T-piece or ventilation with minimal support (pressure support level < 10 cm H2O) and FiO2 ≤ 0.4. In case SBTs are used, an SBT is judged as successful when the following criteria are met for at least 30 minutes, the attending physician takes the final decision for extubation:

* Respiratory rate < 35/min
* Peripheral oxygen saturation > 90%
* Increase < 20% of heart rate and blood pressure
* No signs of anxiety and diaphoresis In case a patient needs to be re-intubated and ventilated, the PEEP level is set as described above.

Sedation follows the local guidelines for sedation in each participating unit. In general, these guidelines favor the use of analgo-sedation over hypno-sedation, use of bolus over continuous infusion of sedating agents, and the use of sedation scores.

Statistical Analysis:

* The statistical analysis will be based on the intention-to-treat principle. In addition, a per-protocol analysis will be performed to check for robustness of results.
* The primary outcome is the number of ventilator-free days and alive at day 28 after ICU admission. The null hypothesis entails that ventilation with the 'restricted PEEP'-arm is inferior by a margin of 10% to ventilation with the 'liberal PEEP'-arm. If the 95% CI upper bound for inferiority of the 'restricted PEEP'-arm is <10%, the null hypothesis of inferiority is rejected. If the non-inferiority criterion is satisfied, then a secondary analysis of the primary endpoint for superiority will be tested. With an appropriate nonparametric analysis method the confidence interval for the difference between the two medians of the ventilator free days from both PEEP arms will be evaluated.
* Continuous normally distributed variables will be expressed by their mean and standard deviation or, when not normally distributed, as medians and their interquartile ranges. Categorical variables will be expressed as frequencies and percentages. Differences between groups in continuous variables will be analyzed with Students t-test or if continuous data is not normally distributed, the Mann-Whitney U test will be used. Categorical variables will be compared with the Chi-squared test or Fisher's exact test, as appropriate. Time-dependent data will be expressed with Kaplan-Meier curves.
* Cost-effectiveness analysis. Alongside the proposed RCT a prospective economic study will be performed. The economic evaluation primarily focuses on the possible gained benefits of ventilation with restricted PEEP versus liberal PEEP and the associated healthcare costs within 28 days (the primary outcome of the RCT). Incremental Cost Effectiveness Ratios (ICER) will be calculated by extra costs per TISS/NAS point, a valuable score reflecting workload and resource utilization in daily ICU practice.
* A budget impact analysis (BIA) will be designed and executed according to the ISPOR guidelines. The BIA will evaluate the nationwide economic/financial consequences of the adoption of treating non-ARDS patients at the ICU with ventilation with restricted PEEP level or liberal PEEP level in the future. The analysis will be based on the decrease in ICU costs (e.g. ventilator free days and alive at day 28) as estimated during the study.

Substudies:

Substudies of the RELAx study ('RELAxECHO', 'RELAxLUS' and 'RELAxBiomarkers') are performed in patients admitted to the ICU of the Academic Medical Center, Amsterdam and who are enrolled in the RELAx study. The protocol of each substudy is described in the appendices of the RELAx protocol: appendix IV 'RELAxECHO'; appendix V 'RELAxLUS' and appendix VI 'RELAxBiomarkers'. The link to the RELAx protocol including the appendices for substudies can be found under 'references'.

Enrolment of RELAx patient in the substudies started on 25th July 2018, 25th July 2018 and 4th December 2018 in the Academic Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating ICUs
* Need for and start of invasive ventilation
* An expected duration of ventilation > 24 hours

Exclusion Criteria:

* Age less than 18 years
* Patients with a clinical diagnosis of ARDS or possible ARDS with a PaO2/FiO2 < 200 mmHg (as the benefit of ventilation with higher PEEP levels has been proven in these patients)
* Patients with ongoing cardiac ischemia due to cardiac infarction and failed revascularization, patients with increased and uncontrollable intracranial pressure (of ≥ 18 mmHg), patients with delayed cerebral ischemia after subarachnoid hemorrhage, patients with necrotizing fasciitis, and severe untreatable anemia such as in case of Jehovah's Witnesses (as these patients can be considered to be vulnerable to the potentially dangerous hypoxemia which could develop more often, even for a short time, in the 'restricted PEEP'-arm of this trial)
* Patients previously randomized in this RCT
* Patients participating in another RCT with the same clinical endpoint, or interventions possibly compromising the primary outcome
* Invasive ventilation longer than 12 hours directly preceding the present ICU admission
* Invasive ventilation longer than 1 hour before randomization
* Patients with suspected or confirmed pregnancy
* Patients with morbid obesity (body mass index > 40)
* Patients with GOLD classification III or IV chronic obstructive pulmonary disease (COPD)
* Patients with premorbid restrictive pulmonary disease (evidence of chronic interstitial infiltration on chest radiographs)
* Patients in whom pulse oximetry is known to be unreliable, e.g., patients with carbon monoxide poisoning
* Any neurologic diagnosis that can prolong duration of mechanical ventilation, e.g., patients with Guillain-Barré syndrome, high spinal cord lesion or amyotrophic lateral sclerosis, multiple sclerosis, or myasthenia gravis
* No informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Ventilation-free days and alive at day 28 | first 28 days after start of ventilation
  The number of ventilation-free days, defined as the number of days from day 1 to day 28; the patient is alive and breathes without assistance of the mechanical ventilator, if the period of unassisted breathing lasted at least 24 consecutive hours.

SECONDARY OUTCOMES:
Length of stay | first 90 days after start of ventilation
  Length of stay in the intensive care unit and in the hospital
Mortality | first 90 days after start of ventilation
  Any death during ICU-, hospital-stay and within 90 days
Pulmonary complications | daily until detubation or day 28
  development of ARDS according tot the Berlin definition, severe hypoxemia, severe atelectasis, severe atelectasis, pneumonia and pneumothorax.
Rescue strategies for severe hypoxemia or severe atelectasis | daily until detubation or day 28
  Recruitment maneuver, prone positioning and bronchoscopy for opening atelectasis.
Days with use of hemodynamic support | daily until detubation or day 28
  The number of ICU days with any use of vasopressors/inotropes for > 2 hours on a day.
Days with use of sedation | daily until detubation or day 28
  Defined as the number of ICU days with any use of sedatives for > 2 hours on a day.
Therapeutic intervention scoring system (TISS)/ Nursing Activities Score (NAS) | daily until detubation or day 28
  Incremental Cost Effectiveness Ratios (ICER) will be calculated by extra costs per TISS/NAS point, a valuable score reflecting workload and resource utilization in daily ICU practice.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J. Schultz, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center; Frederique Paulus, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center
Locations (13):
- Netherlands (13):
  - Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - VU Medical Center, Amsterdam
  - Gelre Hospital, Apeldoorn
  - Rijnstate, Arnhem
  - Amphia Hospital, Breda
  - Spaarne Gasthuis, Hoofddorp
  - Westfriesgasthuis, Hoorn
  - Maastricht University Medical Center, Maastricht
  - Sint Antonius Hospital, Nieuwegein
  - Haaglanden Medical Center, The Hague
  - HagaZiekenhuis, The Hague
  - Isala Clinics, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Meenen DMP, Algera AG, Schuijt MTU, Simonis FD, van der Hoeven SM, Neto AS, Abreu MG, Pelosi P, Paulus F, Schultz MJ; for the NEBULAE; PReVENT; RELAx investigators. Effect of mechanical power on mortality in invasively ventilated ICU patients without the acute respiratory distress syndrome: An analysis of three randomised clinical trials. Eur J Anaesthesiol. 2023 Jan 1;40(1):21-28. doi: 10.1097/EJA.0000000000001778. Epub 2022 Nov 18. PMID 36398740
- [Derived] Writing Committee and Steering Committee for the RELAx Collaborative Group; Algera AG, Pisani L, Serpa Neto A, den Boer SS, Bosch FFH, Bruin K, Klooster PM, Van der Meer NJM, Nowitzky RO, Purmer IM, Slabbekoorn M, Spronk PE, van Vliet J, Weenink JJ, Gama de Abreu M, Pelosi P, Schultz MJ, Paulus F. Effect of a Lower vs Higher Positive End-Expiratory Pressure Strategy on Ventilator-Free Days in ICU Patients Without ARDS: A Randomized Clinical Trial. JAMA. 2020 Dec 22;324(24):2509-2520. doi: 10.1001/jama.2020.23517. PMID 33295981
- [Derived] Algera AG, Pisani L, Bergmans DCJ, den Boer S, de Borgie CAJ, Bosch FH, Bruin K, Cherpanath TG, Determann RM, Dondorp AM, Dongelmans DA, Endeman H, Haringman JJ, Horn J, Juffermans NP, van Meenen DM, van der Meer NJ, Merkus MP, Moeniralam HS, Purmer I, Tuinman PR, Slabbekoorn M, Spronk PE, Vlaar APJ, Gama de Abreu M, Pelosi P, Serpa Neto A, Schultz MJ, Paulus F; RELAx Investigators and the PROVE Network Investigators. RELAx - REstricted versus Liberal positive end-expiratory pressure in patients without ARDS: protocol for a randomized controlled trial. Trials. 2018 May 9;19(1):272. doi: 10.1186/s13063-018-2640-5. PMID 29739430
- See also: RELAx website, link to the study protocol — https://sites.google.com/view/relaxtrial/study-details-and-documents/protocol
- Available data/document: Study Protocol — https://sites.google.com/view/relaxtrial/study-details-and-documents/protocol

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT03167580/SAP_000.pdf
  • Study Protocol (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03167580/Prot_001.pdf